CLINICAL TRIAL: NCT01713777
Title: Equivalence Among Antiepileptic Drug Generic and Brand Products in People With Epilepsy: Chronic-Dose 4-Period Replicate Design (EQUIGEN Chronic-Dose Study)
Brief Title: Equivalence Among Antiepileptic Drug Generic and Brand Products in People With Epilepsy: Chronic-Dose 4-Period Replicate Design
Acronym: Chronic Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Epilepsy Foundation (Other); American Epilepsy Society (Other)
Responsible Party: Principal Investigator, Michael Privitera, Professor, Director Cincinnati Epilepsy Center, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EQUIGEN Chronic Dose; Epilepsy Foundation (Other Grant/Funding Number: 005-1005)
Record Dates: First submitted 2012-10-10; First posted 2012-10-25 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Epilepsy
Keywords: Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamotrigine Generic "A"/Generic "B" (Experimental): Crossover trial. Each arm will receive generic "A" for two periods and generic "B" for two periods.
  Interventions: Drug: Lamotrigine Generic "A"; Drug: Lamotrigine generic "B"
- Lamotrigine Generic "B"/Generic "A" (Experimental): Crossover trial. Each participant will have two periods of generic "A" and two periods of generic "B"
  Interventions: Drug: Lamotrigine Generic "A"; Drug: Lamotrigine generic "B"

INTERVENTIONS:
Drug: Lamotrigine Generic "A"
Drug: Lamotrigine generic "B"

SUMMARY:
The United States Food and Drug Administration (FDA) has specific rules generic drug companies must follow to get a generic copy of a seizure medication approved. Currently, the FDA approves generic drugs by requiring studies on normal volunteers who don't have epilepsy and who take just one dose of the generic drug followed by a series of blood tests. Some people with epilepsy and their physicians have complained about side effects or loss of seizure control when taking generic drugs, but no one knows if these complaints are truly because of problems with the generic drugs.

When the FDA tests generic copies of lamotrigine (LTG), the blood levels measured after volunteers receive the generic lamotrigine tablets are allowed to fall within a specific range. This research will test whether two different manufacturer's generic lamotrigine, that fall in different parts of that range, perform in a similar way when given to people with epilepsy every day over a several week period. The two products will be called GENERIC A and GENERIC B.

The generic forms of the study drug lamotrigine to be tested in this study are approved by the FDA for the treatment of seizures.

DETAILED DESCRIPTION:
Qualified subjects will be screened and upon fulfilling inclusion/exclusion criteria and signing the informed consent will be enrolled into the study and enter the randomization phase (2-30 days). Subjects will be randomized according to a sealed allocation list that will be balanced for sequence and provided to each site prior to the first subject enrollment. Subjects that withdraw prior to completing the second period will be replaced in a randomized manner. The randomization list will be generated by the study statistical group. There are four test periods in two sequences for a sequence-randomized study. During two test periods subjects will receive twice daily dosing of the "low" generic product and during the other two periods subjects will receive twice daily dosing of the "high" generic product. Each subject will return at the end of the 14+/-1 day stable dosing period for an in-facility 12-hour pharmacokinetic (PK) session to collect samples to determine Cmax and AUCs (area under curve). Each in-facility pharmacokinetic testing will be separated by a 14+/-1 day stable dosing period. A final follow-up phone evaluation will be conducted 12-16 days (target 14 days) after the last dose of study medication. A single make-up period will be permitted if there are issues during any single period. During the study the subjects will continue their usual concomitant medications, including AEDs (anti epilepsy drugs), without change.

Investigators will compare the AED levels as measured by Cmax and AUC in each group using average bioequivalence (ABE) and individual bioequivalence (IBE) criteria. Average bioequivalence will be established if the 90% confidence intervals of the geometric mean of Cmax and AUCs for the most disparate generic products compared to each other are entirely within the 80%-125% range (the FDA criteria for bioequivalence) using the two one-sided standard analyses. Otherwise the products will be considered to not be bioequivalent.

Study Population: Approximately 36 subjects (30 subjects to completion).

Number of centers: 3 sites enrolling approximately 12 subjects each.

Duration of study: Approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must satisfy the criteria below at the time of enrollment:

1. 18 years or older.
2. BMI not less than 18.5 and weight not less than 110 pounds.
3. Not donated blood within 56 days of the first pharmacokinetic testing.
4. Agrees not to donate blood at any time during the trial and for 56 days after the final PK in-facility admission.
5. Has had epilepsy for at least one year based on site PIs assessment.
6. Receiving conventional (not extended release) lamotrigine as an antiepileptic drug in twice daily dosing at either 100 mg twice per day, 200 mg twice per day, 300 mg twice per day, or 400 mg twice per day.
7. No changes in AED regimen (lamotrigine or concomitant AED) for at least 28 days prior to first pharmacokinetic testing.
8. Have the ability to understand the informed consent form and be willing to provide informed consent.
9. Willing to remain on same AED regimen through entire study. Subjects will be responsible to supply all of their concomitant medications (except for the study medication, lamotrigine).
10. Willing to stay approximately 14 hours in the research facility on four separate occasions for pharmacokinetic testing.
11. Willing to fast overnight and the morning of each of the four pharmacokinetic testing sessions.
12. Willing to have at least 21 blood samples collected during the pharmacokinetic testing including the in-facility session and outpatient portion for each period. The in-facility blood collections will mainly be performed using an inserted catheter. In the event of difficulty with the catheter or by subject preference, samples may be drawn by venipuncture. The outpatient portion consists of morning trough levels within +/-1 hour of the morning scheduled dose time on the 2 days prior to each research facility PK admission drawn by venipuncture for each of the 4 periods. The total amount of blood during each PK session will be equal to about 12 teaspoons (58.5 milliliters). The total amount of blood drawn throughout the entire study will be about 62 teaspoons (309.5 milliliters) or less. For reference, this amount is approximately two-thirds of the quantity of blood drawn during a standard blood donation by the Red Cross.
13. Willing to completely abstain from alcohol consumption for at least 72-hours prior to each PK in-facility admission (that is from 1 day prior to the first outpatient steady state level) until after the last sample is drawn for each period. Investigators encourage no or minimal alcohol use throughout the study, but alcohol is not restricted at other times.
14. Willing to remain on a consistent regimen of concomitant medications including over-the-counter drugs and herbal drugs, if they are being used and deemed to possibly affect the metabolism of the study medication.
15. Willing to not eat grapefruit or drink grapefruit juice through the duration of the study.
16. If a tobacco user, willing to continue with the same pattern of tobacco use except that no tobacco use is permitted during the PK facility admissions of approximately 14 hours (includes all tobacco products).
17. Willing to complete the subject diary as outlined in the protocol.
18. Willing to adhere to all other protocol requirements as outlined in the informed consent document.
19. Females must be either of non-childbearing potential (defined as having undergone surgical sterilization or postmenopausal (greater than 50 years old and amenorrhea for greater than or equal to 12 months) or must be using at least one acceptable method of contraception as follows:

    1. Double-barrier method (e.g. condom plus spermicide, condom plus diaphragm with spermicide)
    2. Hormonal contraceptive treatment (progesterone only agents - use of any agents containing estrogen are an exclusion for the lamotrigine testing)
    3. Intrauterine Device (IUD)
    4. Monogamous relationship with a vasectomized partner
    5. Abstinent for 8 weeks prior to and throughout the study.
20. Subject must be at least 28 days from last participation in any other study.

Exclusion Criteria:

* 1. Use of an extended release formulation of LTG within 28 days of study entry. 2. Subject is receiving LTG at a total daily dose above 800 mg per day within 28 days of study entry.

  3. Progressive CNS disorder that could influence adverse effects or seizure control.

  4. Known medication non-adherence. Non-adherence is assessed by the investigator based on the procedures defined in the manual of procedures.

  5. Use of valproate (as divalproex sodium or valproic acid), any form of estrogens, rifampin, orlistat, felbamate or sertraline within 28 days of study entry.

  6. Subject has a history of alcohol or substance abuse within 1 year prior to screening of study participation, or is currently using alcohol, drugs of abuse, or any prescribed or over-the-counter medication in a manner, which, in the opinion of the Investigator, indicates abuse.

  7. History of psychogenic seizures within the past 2 years. 8. Any clinically significant psychiatric illness or psychological or behavioral problem which, in the opinion of the investigator, could interfere with the subject being able to participate in the study or comply with the study requirements.

  9. Any clinically significant laboratory abnormality or illness which, in the opinion of the investigator, could interfere with the conduct or interpretation of the study or put the subject at risk.

  10. Pregnant or lactating within 56 days of enrollment. 11. Unstable seizure control that makes AED changes likely during the course of the study.

  12. Use of rescue AEDs (e.g. benzodiazepines) during more than two weeks of the 2 months prior to enrollment.

  13. Subject is in the process of quitting smoking within 28 days of study entry or plans to quit smoking during the period of time the study will be conducted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence for generic 1 compared to generic 2 | 18 months
  To determine if Cmax or AUC are significantly different in the high generic product compared to the low generic product taking one as the reference and the other as the test product. Bioequivalence will be established per the current FDA ABE criteria if the 90% confidence interval of the geometric mean of Cmax and AUC for the high generic product compared to the low generic product are entirely within the 80%-125% range using the two one-sided standard analyses

SECONDARY OUTCOMES:
Intra-subject variances | 18 months
  To measure the intra-subject variances of the investigated generic products, as well as subject-by-interaction variances, by using two replicate periods for each generic product. These estimated variances will be used to investigate individual bioequivalence and detect subject-by-formulation interaction outliers

OTHER OUTCOMES:
Individual Bioequivalence | 18 months
  To examine individual bioequivalence by comparing the two generic products. Individual bioequivalence (IBE) will be determined using the FDA 2001 guidance criteria. To determine the number of subjects who are outliers and to identify these subjects for potential further study.
Bioequivalence for subjects receiving inducers compared to not receiving inducers | 18 months
  To compare the generic1/generic2 ratios for Cmax and AUC in subjects on a concomitant enzyme inducing AED compared to subjects not on a concomitant enzyme AED
Bioequivalence by gender | 18 months
  To compare the generic1/generic2 ratios for Cmax and AUC male subjects compared to female subjects
Bioequivalence in enriched population | 18 months
  To compare the generic1/generic2 ratios for Cmax and AUC in the population of subjects who had reported loss of seizure control or unanticipated adverse effects after a generic switch

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Privitera, MD, Principal Investigator — University of Cincinnati; Michel J Berg, MD, Principal Investigator — University of Rochester
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Drake University, Des Moines, Iowa
  - University of Kansas, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michel J. Berg, MD, Rochester, New York
  - Michael Privitera, MD, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Privitera MD, Welty TE, Gidal BE, Diaz FJ, Krebill R, Szaflarski JP, Dworetzky BA, Pollard JR, Elder EJ Jr, Jiang W, Jiang X, Berg M. Generic-to-generic lamotrigine switches in people with epilepsy: the randomised controlled EQUIGEN trial. Lancet Neurol. 2016 Apr;15(4):365-72. doi: 10.1016/S1474-4422(16)00014-4. Epub 2016 Feb 12. PMID 26875743